CLINICAL TRIAL: NCT07259291
Title: Minto and Eleveld Remifentanil Target Controlled Infusion (TCI) Models: a Clinical Comparison Through qNOX and ANIi Reactions to Post-tetanic Count
Brief Title: Minto and Eleveld Remifentanil Target Controlled Infusion (TCI) Models: a Clinical Comparison
Acronym: TCI
Status: Recruiting | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, PhD, Principal investigator, University of Padova
Other Study IDs: RemiMAST
Record Dates: First submitted 2025-09-29; First posted 2025-12-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Propofol; Anesthesia Brain Monitoring; Remifentanil
Keywords: Analgesia monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eleveld TCI: Patients who received general anesthesia with Eleveld TCI model for Propofol and Remifentanil (this model was choosen at anesthesiologist's discretion)
- Minto TCI: Patients who received general anesthesia with Eleveld TCI model for Propofol and Minto TCI for Remifentanil (this model was choosen at anesthesiologist's discretion)

SUMMARY:
Remifentanil is commonly used as an opioid during general anesthesia. In recent years, several pharmacokinetic/pharmacodynamic (PK/PD) models for target-controlled infusion (TCI) have been developed, with the Eleveld model being one of the most recent and designed for broad applicability.

The aim of this study is to compare the Eleveld TCI model with the routinely used Minto model, in order to evaluate potential differences in the predicted effect-site concentrations (CeR) required to achieve equivalent analgesia levels, as measured by qNOX (CONOX monitor) and the Analgesia Nociception Index (ANI). Post-Tetanic Count (PTC) was also assessed during the maintenance phase to investigate possible differences in nociceptive index responses between the two TCI models.

DETAILED DESCRIPTION:
Remifentanil is a short-acting synthetic opioid frequently used as part of balanced general anesthesia due to its favorable pharmacokinetic profile, which includes rapid onset, short context-sensitive half-time, and predictable elimination. These properties make it ideal for administration via target-controlled infusion (TCI), allowing anesthesiologists to maintain a desired effect-site concentration (Ce) with high precision.

Over the past two decades, several pharmacokinetic/pharmacodynamic (PK/PD) models have been developed to guide TCI of remifentanil. Among these, the Minto model has been widely adopted in routine clinical practice. It was originally derived from data collected in healthy volunteers and incorporates covariates such as age, weight, height, and sex. However, its applicability across broader patient populations has been questioned, particularly in individuals outside the demographic or physiological range of the original dataset.

More recently, the Eleveld model has been introduced as a general-purpose model for remifentanil TCI. It was developed using a large pooled dataset covering a wide range of patient types, including pediatric, adult, and elderly individuals. This model aims to offer more accurate and consistent predictions of drug concentrations and effects across diverse clinical scenarios.

The primary aim of this study is to compare the Eleveld and Minto models with respect to the effect-site concentration (CeR) of remifentanil required to achieve comparable levels of intraoperative analgesia. Analgesia was assessed using two objective nociception monitors: the qNOX index (derived from the CONOX monitor) and the Analgesia Nociception Index (ANI). These indices provide continuous, real-time information on the balance between nociceptive stimulation and the analgesic effect, allowing for a quantitative comparison between the two models.

To further explore the analgesic efficacy and responsiveness under each model, investigators introduced controlled nociceptive stimuli during the maintenance phase of anesthesia. Specifically, the Post-Tetanic Count (PTC) stimulation was applied during anesthesia maintenance to serve as a standardized noxious input. The response of the analgesia monitoring indices (qNOX and ANI) to this stimulus was analyzed, enabling the assessment of how each TCI model modulates analgesic depth in the face of a defined nociceptive challenge.

By comparing the CeR values, the baseline and post-stimulus nociception indices, and their temporal patterns under the two models, this study aims to determine whether the Eleveld model offers any clinical or pharmacodynamic advantages over the traditional Minto model in guiding remifentanil administration during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Undergo general anaesthesia with Targeted Controlled Infusion of Propofol (Eleveld model) and Remifentanil (Minto or Eleveld model)

Exclusion Criteria:

* Neurological disease
* Psychiatric disease

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women undergoing brast cancer surgery with general anesthesia with Propofol and Remifentanil TCI, will be recruited
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Comparison between Concentration at the effector site of Remifentanil (CeR) during anesthesia maintenance | We will consider CeR, qNOX and ANI values during the periprocedural phase
  Discover if there are differences between CeR of Eleveld and Minto TCI to aim at the same analgesic depth as measured by qNOX (40-60) and ANI (50-70)

SECONDARY OUTCOMES:
Comparison between qNOX and ANI reaction to noxious stimulation delivered by Post-tetanic count during maintenance of anesthesia | qNOX, ANIi will be recorded during the periprocedural phase
  Discover if there is indices increase (for qNOX) or decrease (for ANIi) after post-tetanic count stimulation during general anesthesia between the Minto and Eleveld TCI model for Remifentanil
Comparing the incidence of Postoperative Delirium (POD) at anesthesia emergence | CAM will be performed in Post Anesthesia Care Unit, 45 minutes after the end of surgery
  Discover if there are different POD rates detected by Confusion Assessment Method (CAM) between Eleveld or Minto TCI models. Higher POD probability with higher CAM scores
Comparing the incidence of pain at anesthesia emergence | NRS will be performed in Post Anesthesia Care Unit, 45 minutes after the end of surgery.
  Discover if there are different Severe pain rates detected by Numeric Rating Scale (NRS) between Eleveld or Minto TCI models.Higher pain with higher NRS scores
Comparing the incidence of cronic pain after 6 months from surgery | NRS will be performed after 6 months from surgery
  Discover if there are different Severe pain rates detected by Numeric Rating Scale (NRS) between Eleveld or Minto TCI models.Higher pain with higher NRS scores

CONTACTS AND LOCATIONS:
Locations (1):
- ULSS2 Marca Trevigiana, Treviso, Italy

IPD SHARING:
Plan to Share IPD: Undecided